# Appendix A Sample informed consent form (SICF)

Title: A phase 1b open label clinical trial to evaluate HIV-1 neutralization antibody breadth in response to HIV gp120 protein vaccine in HIV-uninfected adults with quiescent Systemic Lupus Erythematosus

HVTN protocol number: HVTN 121

Site: [Insert site name]

Thank you for your interest in our research study. Please read this consent form or ask someone to read it to you. If you decide to join the study, we will ask you to sign or make your mark on this form. We will offer you a copy to keep. We will ask you questions to see if we have explained everything clearly. You can also ask us questions about the study.

Research is not the same as treatment or medical care. The purpose of a research study is to answer scientific questions.

## **About the study**

The HIV Vaccine Trials Network (HVTN) and [Insert site name] are doing a study to test an HIV vaccine given to people who have Systemic Lupus Erythematosus (SLE). Some people may just call this "Lupus." HIV is the virus that causes AIDS. Vaccines against HIV are designed to teach the body to produce antibodies against HIV. Antibodies are one of the body's natural ways of protecting against infections.

People who have Lupus may have immune responses that are unique. The responses might be different from people who do not have Lupus. One of these responses is the body's ability to develop antibodies in response to infections.

Special antibodies called broadly neutralizing antibodies (bnAbs) are able to protect against many different types of an infection, such as the different types of HIV found around the world. Because bnAbs are an important focus of HIV vaccine research, researchers would like to understand more about this immune response in people who have Lupus. They want to better understand how the bnAb responses differ from people who do not have Lupus.

About 16 people will take part in this study at multiple sites. The researcher in charge of this study at this clinic is [Insert name of site PI]. The US National Institutes of Health (NIH) is paying for the study.

### 1. We are doing this study to answer several questions.

How do the immune systems of people with Lupus respond to the study vaccine? (Your immune system protects you from disease.)

- Do the immune systems of people with Lupus make bnAbs in response to the study vaccine?
- Is the study vaccine safe to give to people without active symptoms of Lupus?
- Are people with Lupus able to take the study vaccine without becoming too uncomfortable?

### 2. The study vaccine cannot give you HIV.

The study vaccine is not made from actual HIV. It is impossible for the study vaccine to give you HIV. Also, it cannot cause you to give HIV to someone else.

# 3. The study vaccine likely will not change your risk of becoming infected with HIV if you are exposed to the virus.

Site: Any change to the following boxed text requires approval from HVTN
Regulatory Affairs at vtn.core.reg@hvtn.org. You can remove the box around the text.

The vaccine has been given to thousands of people in other studies. In those studies, most people were not protected from infection with HIV. It's very important to avoid exposure to HIV during and after the study. We will tell you how to avoid HIV.

### 4. This study vaccine is experimental.

The study vaccine is called AIDSVAX® B/E. From here on, we will call it the study vaccine. It is an experimental HIV vaccine. This vaccine is used only in research studies.

The vaccine is being provided by Global Solutions for Infectious Diseases (GSID). The AIDSVAX® B/E vaccine is made of man-made proteins that are similar to proteins from the outer surface of the HIV virus. The vaccine is also made with an adjuvant called aluminum hydroxide. An adjuvant is something added to the vaccine to help the immune system respond better. Aluminum hydroxide adjuvants are used in many licensed vaccines that have been given to millions of people. Your body's immune system may respond to this study vaccine by making antibodies that recognize and fight against HIV proteins. Antibodies are special proteins made by the body that can recognize and prevent infections. The AIDSVAX® B/E vaccine has been given to over 10,000 participants in different studies with people who do not have Lupus.

General risks of vaccines:

Generally, vaccinations are considered safe for people with inactive Lupus.

All vaccines can cause fever, chills, rash, aches and pains, nausea, headache, dizziness, and feeling tired. Vaccines can also cause pain, redness, swelling, or

itching where you got the injection. Most people can still do their planned activities after getting a vaccine. Rarely, people have side effects that limit their normal activities or make them go to the doctor.

Rarely, a vaccine can cause an allergic reaction, including a rash, hives, or trouble breathing. Allergic reactions can be life-threatening. You should tell us if you have ever had a bad reaction to any injection or vaccine.

Very rarely, a vaccine causes an autoimmune disease in a person, or makes an autoimmune disease worse. An autoimmune disease happens when your immune system attacks your own body, instead of attacking an infection. You already have one autoimmune disease, Lupus. We do not know if getting the study vaccine could put you at risk for getting additional autoimmune diseases.

We do not know if getting the study vaccine could impact your Lupus, causing it to flare up. If you have a significant lupus flare up, we will stop your vaccinations and continue to check on your health. We will work with your doctor to get you the care you need.

Risks of the study vaccine:

This section lists the side effects we know about. There may be others that we don't yet know about, even serious ones. We will tell you if we learn about any new side effects.

This AIDSVAX® B/E vaccine has been given to thousands of people who do not have Lupus. The most common symptoms at the injection site were pain and tenderness. In some cases, this resulted in some limited arm movement which went away on its own within a few days. Less often, some people had injection site hardness. The most common reactions in the body were headaches, swollen glands, and muscle or joint aches. Some people also reported feeling weak or having low energy.

A few people had changes in blood and urine test results following injections. We do not know if these changes were caused by the study vaccine. The changes did not cause health problems.

One person experienced a serious allergic reaction immediately after a vaccination with AIDSVAX® B/E. The person was treated and recovered completely in a few hours.

We do not know if participants with Lupus in this study will have similar side effects to those seen in earlier studies with participants who did not have Lupus. Also, people with Lupus may have different side effects.

### Joining the study

### 5. It is completely up to you whether or not to join the study.

Take your time in deciding. If it helps, talk to people you trust, such as your doctor, friends or family. If you decide not to join this study, or if you leave it after you have joined, your other care at this clinic and the benefits or rights you would normally have will not be affected.

If you join this study, you may not be allowed to join other HIV vaccine or HIV prevention studies now or in the future. You cannot be in this study while you are in another study where you get a study product. Being in more than one study may not be safe.

Also during the study, you should not donate blood or tissue.

If you choose not to join this study, you may be able to join another study.

Site: Remove item 6 if you use a separate screening consent that covers these procedures.

### 6. If you want to join the study, we will screen you to see if you are eligible.

Screening involves a physical exam, HIV test and health history. A physical exam may include, but is not limited to:

- Checking your weight, temperature and blood pressure
- Looking in your mouth and throat
- Listening to your heart and lungs
- Feeling your abdomen (stomach and liver)

We will also do blood and urine tests. These tests tell us about some aspects of your health, such as how healthy your kidneys, liver, and immune system are, and if you have diabetes. We will also test you for: Syphilis, Hepatitis B, and Hepatitis C. We will ask you about medications you are taking. We will ask you about behaviors that might put you at risk for getting HIV. If you were assigned female sex at birth, we will test you for pregnancy.

We will assess your Lupus status to see if you have any currently active symptoms. This includes blood tests, a physical exam, and a questionnaire.

We may need to review your medical records. We will ask for your permission if this is needed.

We will review the screening results with you. The screening results may show you are not eligible to join the study, even if you want to.

Site: Adapt the following section so it is applicable to the care available at your site

7. If we find that you have a health problem during screening or during the study, we will tell you about the care that we can give here.

For the care that we cannot give, we will explain how we will help you get care elsewhere. For health problems that are unrelated to the study, we will not pay for care.

8. If you were assigned female sex at birth and could become pregnant, you must agree to use birth control to join this study.

Site: If you want to include Appendix B, Approved birth control methods (for sample informed consent form), in this consent form, paste it below and delete paragraph below.

You should not become pregnant during the study because we do not know how the study vaccine could affect the developing baby. You must agree to use effective birth control from 21 days before your first injection until after your last required protocol clinic visit. We will talk to you about effective birth control methods. They are listed on a handout that we will give to you.

## Being in the study

If you meet the study requirements and want to join, here is what will happen:

9. You will come to the clinic for scheduled visits about [#] times over 12 months.

Site: Insert number of visits and range of visit lengths. (There is site-specific variation in screening protocols and in the number of possible follow-up visits between protocol-mandated visits.)

Visits can last from [#] to [#] hours.

You may have to come for more visits if you have a lab or health issue.

We may contact you after the study ends (for example, to tell you about the study results).

10. We will give you [Site: Insert compensation] for each study visit you complete.

This amount is to cover the costs of [Site: Insert text]

Site: Insert any costs to participants (eg, birth control costs for female participants who could become pregnant).

Site: Include the following paragraph. You can remove the box around the text.

Payments you receive for being in the study may be taxable. We may need to ask you for your Social Security number for tax reasons.

You do not have to pay anything to be in this study. The study vaccine, the medical visits, and laboratory tests related to this study will be covered by the clinic, through the study sponsor. However, routine medical care (care you would have received whether or not you were in this study) will be charged to you or your insurance company. You may wish to contact your insurance company to discuss this further.

### 11. We will give you the study product on a schedule.

You will get 3 injections during the study by injection into the muscle of your upper arm.

| Injection schedule | | |
|-------------------------|--------------|--------------|
| First vaccination visit | 1 month | 6 months |
| AIDSVAX® B/E | AIDSVAX® B/E | AIDSVAX® B/E |

You will have to wait in the clinic for about a half hour after each injection to see if there are any problems. Then for that night and for 7 more days, you will need to keep track of how you are feeling and if you have any symptoms. Within 3 days of each injection, we will also ask you how you are doing. Contact the clinic staff if you have any issues or concerns after getting an injection. If you have a problem, we will continue to check on you until it goes away.

### 12. In addition to giving you the study product, we will:

- Do regular HIV testing, as well as counseling on your results and on how to avoid getting HIV
- Do physical exams
- Do pregnancy tests if you were assigned female sex at birth
- Ask questions about your health, including medications you may be taking
- Ask questions about any personal problems or benefits you may have from being in the study
- Assess your Lupus status

• Take urine and blood samples.

When we take blood, the amount will depend on the lab tests we need to do. It will be some amount between 15 mL and 315 mL (1 tablespoon to  $1\frac{1}{2}$  cups). Your body will make new blood to replace the blood we take out.

Site: You may want to add a sentence to the end of the previous paragraph contextualizing the blood volumes described (eg, "To compare, people who donate blood in the US can give a total of about 500 mL in an 8-week period."). Modify the example for cultural relevance and alter blood volumes as necessary.

Site: Insert Appendix D, Table of procedures (for informed consent form) in this section or distribute it as a separate sheet if it is helpful to your study participants. You are not required to do either.

We will be looking for side effects. We will review the results of these procedures and tests with you at your next visit, or sooner if necessary. If any of the results are important to your health, we will tell you.

It is important that you contact the clinic if you have any symptoms between your vaccination and the next scheduled visit. If you think you are having a flare up, please contact the clinic as soon as possible.

### 13. We will counsel you on avoiding HIV infection.

We will ask you personal questions about your HIV risk factors such as sexual behavior, alcohol, and drug use. We will talk with you about ways to keep your risk of getting HIV low.

# 14. The HVTN will test your samples to see how your immune system responds to the study product.

We will send your samples (without your name) to labs approved by the HVTN for this study, which are located in the United States. In rare cases, some of your samples may be sent to labs approved by the HVTN in other countries for research related to this study.

Researchers may also do genetic testing related to this study on your samples. Your genes are passed to you from your birth parents. They affect how you look and how your body works. The differences in people's genes can help explain why some people get a disease while others do not. The genetic testing will only involve some of your genes, not all of your genes (your genome). The researchers will study only the genes related to the immune system and HIV and those that affect how people get HIV.

If you become HIV infected, the researchers may look at all of the genes of the virus found in your samples. The researchers will use this information to learn more about HIV and the study product.

In some cases, researchers may take cells from your samples and grow more of them over time, so that they can continue to contribute to this study.

These tests done on your samples are for research purposes, not to check your health. The labs will not give the results to you or this clinic because their tests are not approved for use in making health care decisions. These labs are only approved to do research tests.

When your samples are no longer needed for this study, the HVTN will continue to store them.

Site: Delete next section if using separate consent for use of samples and information in other studies

# 15. When samples are no longer needed for this study, the HVTN wants to use them in other studies and share them with other researchers.

The HVTN calls these samples "extra samples". The HVTN will only allow your extra samples to be used in other studies if you agree to this. You will mark your decision at the end of this form. If you have any questions, please ask.

Do I have to agree? No. You are free to say yes or no, or to change your mind after you sign this form. At your request, we will destroy all extra samples that we have. Your decision will not affect your being in this study or have any negative consequences here.

Where are the samples stored? Extra samples are stored in a secure central place called a repository. Your samples will be stored in the HVTN repository in the United States.

How long will the samples be stored? There is no limit on how long your extra samples will be stored. [Site: Revise the previous sentence to insert limits if your regulatory authority imposes them.]

Will I be paid for the use of my samples? No. Also, a researcher may make a new scientific discovery or product based on the use of your samples. If this happens, there is no plan to share any money with you. The researcher is not likely to ever know who you are.

Will I benefit from allowing my samples to be used in other studies? Probably not. Results from these other studies are not given to you, this clinic, or your doctor. They are not part of your medical record. The studies are only being done for research purposes.

Will the HVTN sell my samples and information? No, but the HVTN may share your samples with HVTN or other researchers. Once we share your samples and information, we may not be able to get them back.

How do other researchers get my samples and information? When a researcher wants to use your samples and information, their research plan must be approved by the HVTN. Also, the researcher's institutional review board (IRB) or ethics committee (EC) will review their plan. [Site: If review by your institution's IRB/EC/RE is also required, insert a sentence stating this.] IRBs/ECs protect the rights and well-being of people in research. If the research plan is approved, the HVTN will send your samples to the researcher's location.

What information is shared with HVTN or other researchers? The samples and information will be labeled with a code number. Your name will not be part of the information. However, some information that we share may be personal, such as your race, ethnicity, sex, health information from the study, and HIV status. We may share information about the study product you received and how your body responded to the study product.

What kind of studies might be done with my extra samples and information? The studies will be related to HIV, vaccines, the immune system and other diseases.

Researchers may also do genetic testing on your samples.

In some cases, researchers may take cells from your samples and grow more of them over time, so that they can continue to do research with them.

If you agree, your samples could also be used for genome-ide studies. In these studies, researchers will look at all of your genes (your genome). The researchers compare the genomes of many people, looking for common patterns of genes that could help them understand diseases. The researchers may put the information from the genome-wide studies into a protected database so that other researchers can access it, but your name and other personal information will not be included. Usually, no one would be able to look at your genome and link it to you as a person. However, if another database exists that also has information on your genome and your name, someone might be able to compare the databases and identify you. If others found out, it could lead to discrimination or other problems. The risk of this is very small. There may be other unknown risks.

Who will have access to my information in studies using my extra samples?

People who may see your information are:

- Researchers who use your extra samples and information for other research
- Government agencies that fund or monitor the research using your extra samples and information
- The researcher's Institutional Review Board or Ethics Committee
- Any regulatory agency that reviews clinical trials

## The people who work with the researcher

All of these people will do their best to protect your information. The results of any new studies that use your extra samples and information may be published. No publication will use your name or identify you personally.

### 16. We will do our best to protect your private information.

Site: Check Health Insurance Portability and Accountability Act (HIPAA) authorization for conflicts with this section.

Your study records and samples will be kept in a secure location. We will label all of your samples and most of your records with a code number, not your name or other personal information. However, it is possible to identify you, if necessary. We will not share your name with the lab that does the tests on your samples, or with anyone else who does not need to know your name.

Site: Any change to the following boxed text requires approval from HVTN Regulatory Affairs. You can remove the box around the text.

We do need to share your name with the HVTN in case you need proof in the future that you participated in an HIV vaccine study. The HVTN will keep your name in a secure file with these items:

- The name of your study
- Your age or date of birth
- Your study ID number
- What study product you received

There are no HIV test results kept in this file. The HVTN will not share any information that could identify you without your agreement. The HVTN will remove your name from the file if you do not want it there.

Clinic staff will have access to your study records. Your records may also be reviewed by groups who watch over this study to see that we are protecting your rights, keeping you safe, and following the study plan. These groups include:

- The US National Institutes of Health (NIH) and its study monitors,
- The US Food and Drug Administration (FDA),
- Any regulatory agency that reviews clinical trials
- [Insert name of local IRB/EC],

- [Insert name of local and/or national regulatory authority as appropriate],
- Global Solutions for Infectious Diseases (GSID) and people who work for them,
- The HVTN and people who work for them,
- The HVTN Safety Monitoring Board, and
- The US Office for Human Research Protections (OHRP).

All reviewers will take steps to keep your records private.

We cannot guarantee absolute privacy. At this clinic, we have to report the following information:

Site: Include any public health or legal reporting requirements. Bulleted examples should include all appropriate cases (reportable communicable disease, risk of harm to self or others, etc.).

- [Item 1]
- [Item 2]
- [Item 3]

Site: Include the following boxed text. You can remove the box around the text.

We have a Certificate of Confidentiality from the US government, to help protect your privacy. With the certificate, we do not have to release information about you to someone who is not connected to the study, such as the courts or police. Sometimes we can't use the certificate. Since the US government funds this research, we cannot withhold information from it. Also, you can still release information about yourself and your study participation to others.

The results of this study may be published. No publication will use your name or identify you personally.

We may share information from the study with other researchers. We will not share your name or information that can identify you.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# 17. We may stop your injections or take you out of the study at any time. We may do this even if you want to stay in the study and even if you were scheduled for more injections.

This may happen if:

- you do not follow instructions,
- we think that staying in the study might harm you,
- you have more than a mild Lupus flare,
- you enroll in a different research study where you get another study product, or
- the study is stopped for any reason.

If we stop your injections, we may ask you to stay in the study to complete other study procedures.

### 18. We will stop your injections if you become pregnant.

We will encourage you to stay in the study if you choose. We will discuss your study options with you.

If you leave the study while you are still pregnant, we will contact you after your due date to ask some questions about your pregnancy and delivery.

# 19. If you get infected with HIV during the study, we will stop your injections, take fewer samples, and help you get care and support.

We will encourage you to stay in the study for up to 24 weeks if you choose. We will discuss your study options with you. We will counsel you about your HIV infection and about telling your partner(s). We will tell you where you can get support and medical care. *Site: Modify the following sentence as appropriate.* We will not provide or pay for any of your HIV care directly.

### Other Risks

### 20. There are other risks to being in this study.

This section describes the other risks and restrictions we know about. There may also be unknown risks, even serious ones. We will tell you if we learn anything new that may affect your willingness to stay in the study.

*Risks of routine medical procedures:* 

In this study, we will do some routine medical procedures. These are taking blood and giving injections. These procedures can cause bruising, pain, fainting, soreness, redness, swelling, itching, a sore, bleeding, and (rarely) muscle damage or infection where you got the injection. Taking blood can cause a low blood cell count (anemia), making you feel tired.

Personal problems/discrimination/testing HIV antibody positive:

About 10 to 20% of people who join HVTN studies report personal problems or discrimination because of joining an HIV vaccine study. Family or friends may worry, get upset or angry, or assume that you are infected with HIV or at high risk and treat you unfairly as a result. Rarely, a person has lost a job because the study took too much time away from work, or because their employer thought they had HIV.

The body makes antibodies to fight or prevent infection. Most vaccines cause the body to make antibodies as a way of preventing infection. Your body may make antibodies to HIV because you received an HIV vaccine. The study vaccine may cause you to test positive on some types of HIV antibody tests, even if you are not infected with HIV. This is called vaccine-induced seropositivity (VISP). VISP means that after you get the study vaccine, a routine HIV test done outside this clinic [may / is likely to] say you have HIV, even if you don't. For this reason, you should plan to get HIV tests only at this clinic during the study. Our tests can tell the difference between true HIV infection and a positive result that is caused by the study vaccine.

If you have a positive test result caused by the study vaccine at any time, we can arrange free HIV testing for as long as you need it. If this happens, we do not know how long you will test positive due to the study vaccine. If you receive a positive HIV test result and we determine it is because you have HIV, we will refer you for follow-up care.

It is unlikely, but you could test negative at the end of the study and positive some time later, even though you don't have HIV. This could happen if different HIV tests come into use. We will give you a phone number to call for more information.

Site: Modify the following paragraph if applicable. If someone believes you are infected with HIV even if you are not, you could face discrimination and other problems. For example, in some countries, you could be denied medical or dental care, employment, insurance, a visa, or entry into the military. If you do have a positive HIV antibody test caused by the study vaccine, you will not be able to donate blood or organs. Your family and friends may treat you differently. We will give you a brochure that tells you more about testing HIV positive because of an HIV vaccine, and how you can avoid some of these problems.

If you become pregnant during or after the study and have VISP, we don't know if the antibodies could be passed to your baby. We know that this happens with other vaccines, like tetanus vaccine. These antibodies from the mother are not a danger to the baby, and they go away over time. For most babies antibodies from the mother last for about six months.

You should always tell the delivery staff if you have VISP. However, you may still be tested for HIV using the antibody test when you deliver your baby. If your test is positive and the delivery staff believes you have an HIV infection, your baby may be started on antiretroviral treatment when it is not needed. If this happens, we can arrange for you and the baby to have a test that can tell the difference between true HIV infection and a VISP result. If you or the baby continue to have VISP, we can arrange this testing for free for as long as it is needed.

### Embarrassment/anxiety:

You may feel embarrassed when we ask about your HIV risks, such as having sex and using drugs. Also, waiting for your HIV test results or other health test results could make you feel anxious. You could feel worried if your test results show that you are infected with HIV. If you feel embarrassed or anxious, please tell us and we will try to help you.

### Risks of disclosure of your personal information:

We will take several steps to protect your personal information. Although the risk is very low, it is possible that your personal information could be given to someone who should not have it. If that happened, you could face discrimination, stress, and embarrassment. We can tell you more about how we will protect your personal information if you would like it.

### Risks of genetic testing:

It is unlikely, but the genetic tests done on your samples could show you may be at risk for certain diseases. If others found out, it could lead to discrimination or other problems. However, it is almost impossible for you or others to know your test results from the genetic testing. The results are not part of your study records and are not given to you.

In the very unlikely event that your genetic information becomes linked to your name, a federal law called the Genetic Information Nondiscrimination Act (GINA) helps protect you. GINA keeps health insurance companies and employers from seeing results of genetic testing when deciding about giving you health insurance or offering you work. GINA does not help or protect you against discrimination by companies that sell life, disability, or long-term care insurance.

#### Unknown risks:

We do not know if the study vaccine will increase, decrease, or not change your risk of becoming infected with HIV if exposed. If you get infected with HIV, we

do not know how the study vaccine might affect your HIV infection or how long it takes to develop AIDS.

We do not know if getting this study vaccine will affect how you respond to any future approved HIV vaccine. Currently, no HIV vaccine has been approved for use.

We do not know how the study vaccine will affect a pregnant participant or a developing baby.

### **Benefits**

### 21. The study may not benefit you.

We do not expect that the study vaccine will benefit you in any way. We do not know if there will be benefit from this research for the larger community of people who have Lupus. However, being in the study might still help you in some ways. The counseling that you get as part of the study may help you avoid getting HIV. The lab tests and physical exams that you get while in this study might detect health problems you don't yet know about.

This study may help in the search for a vaccine to prevent HIV. The information learned in this study will help to inform the larger field of HIV vaccine research. However, if the study vaccine later becomes approved and sold, there are no plans to share any money with you.

## Your rights and responsibilities

### 22. If you join the study, you have rights and responsibilities.

You have many rights that we will respect. You also have responsibilities. We list these in the Participant's Bill of Rights and Responsibilities. We will give you a copy of it.

# Leaving the study

### 23. Tell us if you decide to leave the study.

You are free to leave the study at any time and for any reason. Your care at this clinic and your legal rights will not be affected, but it is important for you to let us know.

We will ask you to come back to the clinic one last time for a physical exam, and we may ask to take some blood and urine samples. We will also ask about any personal problems or benefits you have experienced from being in the study. We believe these steps are important to protecting your health, but it is up to you whether to complete them.

### Injuries

Site: Approval from HVTN Regulatory Affairs (at vtn.core.reg@hvtn.org) is needed for any change (other than those that the instructions specifically request or those previously approved by HVTN Regulatory Affairs) to the boxed text. You can remove the box around the text.

### 24. If you get sick or injured during the study, contact us immediately.

Your health is important to us. (Site: Adjust the following 2 sentences if applicable to the care available at your site) We will tell you about the care that we can give here. For the care that we cannot provide, we will help you get care elsewhere by referring you for treatment.

If you become sick or injured in this study, please tell your study doctor. There are no funds to pay for treatment of study-related injuries or Lupus flares (regardless of whether or not they are study related). Your insurance company may not be willing to pay for study-related injury or for Lupus flares that occur while you are in the study. If you have no insurance, you would be responsible for any costs.

### Questions

25. If you have questions or problems at any time during your participation in this study, use the following important contacts.

If you have questions about this study, contact [name or title and telephone number of the investigator or other study staff].

If you have any symptoms that you think may be related to this study, contact [name or title and telephone number of the investigator or other study staff].

This study has been reviewed and approved by a committee called the [name of local IRB/EC]. If you have questions about your rights as a research participant, or problems or concerns about how you are being treated in this study, contact [name or title and telephone number of person on IRB/EC], at the committee.

If you want to leave this study, contact [name or title and telephone number of the investigator or other study staff].

## Your permissions and signature

Site: Delete this section if using a separate consent for use of samples and information in other studies

26. In Section 14 of this form, we told you about possible other uses of your extra samples and information, outside this study. Please choose only one of the

options below and write your initials or make your mark in the box next to it. Whatever you choose, the HVTN keeps track of your decision about how your samples and information can be used. You can change your mind after signing this form.

| Clinic staff conduction discussion ( | | Clinic staff signature | Date | Time |
|---|---|---|---|---|
| Participant's na | me (print) | Participant's signature or mark | Date | Time |
| You wil | ll not be giving up | o any of your rights by signing the | is consent form | n. |
| • You | agree to join this | study. | | |
| • You | have had your qu | uestions answered and know that | you can ask m | nore. |
| | | lerstand what the study is about a understand what the possible risk | | |
| • You | have read this co | onsent form, or someone has read | it to you. | |
| below. | • | study, you will need to sign or not be make your mark on this cons | - | |
| | _ | extra samples to be used in any oth<br>testing, growing more of my cells, o | | |
| OR | | | | |
| | | agree to the option above <i>and</i> also to allow my extra samples and information to be sed in genome wide studies. | | |
| OR | | | | |
| | vaccines, the imm | samples and information to be used to<br>nune system, and other diseases. Thi<br>growing over time. | | |

For participants who are unable to read or write, a witness should complete the signature block below:

Witness's name (print) Witness's signature Date Time

\*Witness is impartial and was present for the entire discussion of this consent form.